CLINICAL TRIAL: NCT01098266
Title: NGR015: Randomized Double-blind Phase III Study of NGR-hTNF Plus Best Investigator's Choice (BIC) Versus Placebo Plus BIC in Previously Treated Patients With Advanced Malignant Pleural Mesothelioma (MPM)
Brief Title: NGR015: Study in Second Line for Patient With Advanced Malignant Pleural Mesothelioma Pretreated With Pemetrexed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGR015; 2009-016879-29 (EudraCT Number)
Record Dates: First submitted 2010-03-17; First posted 2010-04-02 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-08

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: MPM; NGR-hTNF; NGR-hTNF plus BIC; Randomized double-blind phase III study
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: NGR-hTNF + BIC (Experimental): NGR-hTNF plus Best Investigator's Choice
  Interventions: Drug: NGR-hTNF plus Best Investigator's Choice (BIC)
- B: Placebo+BIC (Placebo Comparator): Placebo plus Best Investigator's Choice
  Interventions: Drug: Placebo plus Best Investigator's Choice (BIC)

INTERVENTIONS:
Drug: NGR-hTNF plus Best Investigator's Choice (BIC) — * NGR-hTNF: 0.8 mcg/m² as 60-minute intravenous infusion every week until confirmed evidence of disease progression or unacceptable toxicity occurs.
  * Best Supportive Care: antibiotics, analgesics, antiemetics, thoracentesis, pleurodesis, blood transfusions, nutritional support, and focal external-beam radiation for control of pain, cough, dyspnea, or hemoptysis
  * Investigator's Choice: one of the following single-agent chemotherapy might be administered in combination:
    1. Doxorubicin: 60-75 mg/m2 every 3 weeks, for a maximum of 6 cycles
    2. Gemcitabine: 1,000-1,250 mg/m2 on days 1 and 8, every 3 weeks, for a maximum of 6 cycles
    3. Vinorelbine: 25 mg/m2 iv (or 60 mg/m2 per os) on days 1 and 8, every 3 weeks, for a maximum of 6 cycles (or weekly for 12 weeks)
  Other Names: NGR-hTNF+BIC
  Arms: A: NGR-hTNF + BIC
Drug: Placebo plus Best Investigator's Choice (BIC) — * Placebo: 0.8 mcg/m² as 60-minute intravenous infusion every week until confirmed evidence of disease progression or unacceptable toxicity occurs.
  * Best Supportive Care: antibiotics, analgesics, antiemetics, thoracentesis, pleurodesis, blood transfusions, nutritional support, and focal external-beam radiation for control of pain, cough, dyspnea, or hemoptysis
  * Investigator's Choice: one of the following single-agent chemotherapy might be administered in combination:
    1. Doxorubicin: 60-75 mg/m2 every 3 weeks, for a maximum of 6 cycles
    2. Gemcitabine: 1,000-1,250 mg/m2 on days 1 and 8, every 3 weeks, for a maximum of 6 cycles
    3. Vinorelbine: 25 mg/m2 iv (or 60 mg/m2 per os) on days 1 and 8, every 3 weeks, for a maximum of 6 cycles (or weekly for 12 weeks)
  Other Names: Placebo+BIC
  Arms: B: Placebo+BIC

SUMMARY:
The main objective of the trial is to document the efficacy of NGR-hTNF administered at low dose weekly in advanced Malignant Pleural Mesothelioma patients previously treated with a pemetrexed-based chemotherapy regimen.

DETAILED DESCRIPTION:
Currently, there are no regulatory-approved or widely accepted treatment options for patients failing a standard pemetrexed-based chemotherapy regimen.

For this reason, the best supportive care (BSC) alone might be considered as a standard reference for a randomized phase III trial in this setting.

However, single-agent chemotherapeutic agents (such as doxorubicin,gemcitabine, or vinorelbine) with a well-documented safety profile and antitumor activity are also used in clinical practice.

Therefore, the best investigator's choice (BIC) between either best supportive care alone or combined with a few selected single-agent chemotherapy (including doxorubicin, gemcitabine, or vinorelbine) might be considered as an acceptable reference arm as well in this setting.

The current phase III study aims to show a superior efficacy in terms of overall survival duration of NGR-hTNF 0.8 µg/mq weekly plus BIC versus placebo plus BIC in advanced MPM patients progressing after a standard pemetrexed-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically or cytological confirmed malignant pleural mesothelioma of any of the following subtype: epithelial, sarcomatoid, mixed, or unknown
* Prior treatment with no more than one systemic pemetrexed-based chemotherapy regimen administered for advanced or metastatic disease. Prior use of a biological agent in combination with a pemetrexed-based regimen and prior administration of intrapleural cytotoxic agents are allowed. Patients who have previously received anthracyclines should not receive doxorubicin
* ECOG Performance Status 0 - 2
* Life expectancy of ≥ 12 weeks
* Adequate baseline bone marrow, hepatic and renal function, defined as follows:

  1. Neutrophils ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L; hemoglobin ≥ 9 g/dL
  2. Bilirubin ≤ 1.5 x ULN
  3. AST and/or ALT ≤ 2.5 x ULN in absence of liver metastasis or ≤ 5 x ULN in presence of liver metastasis
  4. Serum creatinine < 1.5 x ULN
* Measurable or non-measurable disease according to MPM-modified RECIST criteria
* Patients may have had prior therapy providing the following conditions are met:

  1. Surgery: wash-out period of 14 days
  2. Systemic and radiation anti-tumor therapy: wash-out period of 28 days
* Patients must give written informed consent to participate in the study

Exclusion Criteria:

* Patients must not receive any other investigational agents while on study
* Patients with myocardial infarction within the last six months, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* Uncontrolled hypertension
* QTc interval (congenital or acquired) > 450 ms
* History or evidence upon physical examination of CNS disease unless adequately treated (e.g., primary brain tumor, any brain metastasis, seizure not controlled with standard medical therapy, or history of stroke)
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Known hypersensitivity/allergic reaction to human albumin preparations or to any of the excipients
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-04-12 (Actual); Primary Completion 2014-04-29 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lambiase, MD, Study Director — AGC Biologics S.p.A.
Locations (49):
- United States (7):
  - Wilshire Oncology Medical Group, Corona, California
  - City of Hope-Comprehensive Cancer Cente, Duarte, California
  - H. Lee Moffitt ancer Center and Research Institute, Tampa, Florida
  - Johns Hopkins, Baltimore, Maryland
  - Columbia University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UTsouthwestern medical center, Dallas, Texas
- Belgium (5):
  - Antwerp University Hospital, Edegem, Antwerp
  - Centre Hospitalier Universitaire de Liège, Liège, Liege
  - Institut Jules Bordet, Brussels
  - Cliniques Universitarie St. Luc, Brussels
  - Universitair Ziekenhuis, Ghent
- Canada (2):
  - UAB - Alberta Cancer Board - Cross Cancer Institute, Edmonton, Alberta
  - University Health Network, Princess Margaret Hospital, Toronto, Ontario
- National Cancer Institute, Cairo, Egypt
- Hôpitaux de Marseille Hôpital Nord, Marseille, France
- St James's Hospital, Dublin, Ireland
- Italy (15):
  - Ospedale Santo Spirito, Casale Monferrato, Alessandria
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano, Torino
  - Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria, Alessandria
  - Centro di Riferimento Oncologico, Aviano
  - Ospedale Valduce, Como
  - Azienda Ospedaliero-Universitaria Careggi di Firenze, Florence
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori-IRST, Meldola
  - Fondazione San Raffaele del Monte Tabor, Milan
  - Azienda Ospedaliera San Gerardo, Monza
  - Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Azienda Unità Sanitaria locale di Ravenna, Ravenna
  - A.O. Salvini Garbagnate, Ospedale di Rho, Rho
  - Azienda Ospedaliera Senese, Siena
- Netherlands (2):
  - St. Jansdal Hospital, Harderwijk, Gelderland
  - St. Antonius Hospital, Nieuwegein, Utrecht
- Poland (2):
  - Medical University of Gdansk, Gdansk
  - Maria Sklodowska Memorial Cancer Center and Institute of Oncology, Warsaw
- Spain (2):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Vall d'Hebron, Barcelona
- The University Hospital, Linköping, Sweden
- United Kingdom (10):
  - Chest Clinic, Wythenshawe Hospital, Manchester, Greater Manchester
  - Kent Oncology Centre Maidstone Hospital, Maidstone, Kent
  - University Hospitals of Leicester, Leicester, Leicestershire
  - Mount Vernon Cancer Centre, Middlesex, Northwood
  - Edinburgh Cancer Centre, Western General Hospital, Edinburgh, Scotland
  - The Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - The Royal Marsden Hospital, Sutton, Surrey
  - Castle Hill Hospital, Cottingham, Yorkshire
  - Guy's Hospital, London
  - The Royal Marsden Hospital, London

REFERENCES:
- [Derived] Gregorc V, Gaafar RM, Favaretto A, Grossi F, Jassem J, Polychronis A, Bidoli P, Tiseo M, Shah R, Taylor P, Novello S, Muzio A, Bearz A, Greillier L, Fontana F, Salini G, Lambiase A, O'Brien M. NGR-hTNF in combination with best investigator choice in previously treated malignant pleural mesothelioma (NGR015): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet Oncol. 2018 Jun;19(6):799-811. doi: 10.1016/S1470-2045(18)30193-1. Epub 2018 May 9. PMID 29753703

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Period: April 12th, 2010(First enrolment); January 21st, 2013 (date of last enrolment); April 29th, 2014 (cut-off date). 15 clinical sites in Italy, 10 in UK, 7 in USA, 4 in Belgium, 2 in Canada, 2 in Netherland, 2 in Poland, 1 in Egypt, 1 in Ireland;1 in Sweden
Pre-assignment Details: Before randomization, the physician had to decide for each patient if he/she was candidate to either Best Supportive Care (BSC) alone or combined with single-agent chemotherapy.
Groups:
- A: NGR-hTNF + BIC: NGR-hTNF plus Best Investigator's Choice
  NGR-hTNF plus Best Investigator's Choice (BIC): - NGR-hTNF: 0.8 mcg/m² as 60-minute intravenous infusion every week until confirmed evidence of disease progression or unacceptable toxicity occurs.
  * Best Supportive Care: antibiotics, analgesics, antiemetics, thoracentesis, pleurodesis, blood transfusions, nutritional support, and focal external-beam radiation for control of pain, cough, dyspnea, or hemoptysis
  * Investigator's Choice: one of the following single-agent chemotherapy might be administered in combination:
    1. Doxorubicin: 60-75 mg/m2 every 3 weeks, for a maximum of 6 cycles
    2. Gemcitabine: 1,000-1,250 mg/m2 on days 1 and 8, every 3 weeks, for a maximum of 6 cycles
    3. Vinorelbine: 25 mg/m2 iv (or 60 mg/m2 per os) on days 1 and 8, every 3 weeks, for a maximum of 6 cycles (or weekly for 12 weeks)
- B: Placebo+BIC: Placebo plus Best Investigator's Choice
  Placebo plus Best Investigator's Choice (BIC): - Placebo: 0.8 mcg/m² as 60-minute intravenous infusion every week until confirmed evidence of disease progression or unacceptable toxicity occurs.
  * Best Supportive Care: antibiotics, analgesics, antiemetics, thoracentesis, pleurodesis, blood transfusions, nutritional support, and focal external-beam radiation for control of pain, cough, dyspnea, or hemoptysis
  * Investigator's Choice: one of the following single-agent chemotherapy might be administered in combination:
    1. Doxorubicin: 60-75 mg/m2 every 3 weeks, for a maximum of 6 cycles
    2. Gemcitabine: 1,000-1,250 mg/m2 on days 1 and 8, every 3 weeks, for a maximum of 6 cycles
    3. Vinorelbine: 25 mg/m2 iv (or 60 mg/m2 per os) on days 1 and 8, every 3 weeks, for a maximum of 6 cycles (or weekly for 12 weeks)
Period: Overall Study
Arm/Group | A: NGR-hTNF + BIC | B: Placebo+BIC
Started | 200 | 200
Completed | 193 | 193
Not Completed | 7 | 7
Not completed — Physician Decision | 1 | 0
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Population: Patients ≥ 18 years with advanced malignant pleural mesothelioma previously treated with a pemetrexed based chemotherapy regimen for advanced or metastatic disease.
Groups:
- Total: Total of all reporting groups
Arm/Group | A: NGR-hTNF + BIC | B: Placebo+BIC | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 92 | 87 | 179
  >=65 years | 108 | 113 | 221
Age, Continuous [Median (Full Range); unit: years] | 65 [25 to 89] | 67 [31 to 81] | 66 [25 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 55 | 99
  Male | 156 | 145 | 301
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 198 | 197 | 395
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 5 | 8
  Netherlands | 5 | 2 | 7
  Sweden | 1 | 1 | 2
  Belgium | 5 | 8 | 13
  United States | 14 | 12 | 26
  Ireland | 3 | 1 | 4
  Egypt | 17 | 19 | 36
  Poland | 17 | 14 | 31
  Italy | 79 | 84 | 163
  United Kingdom | 49 | 46 | 95
  France | 4 | 6 | 10
  Spain | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Defined as the time from the date of randomization until the date of death due to any cause or the last date the patient was known to be alive
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, wichever came first, assesed up to 48 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A: NGR-hTNF + BIC | B: Placebo+BIC
Number analyzed (Participants) | 200 | 200
months | 8.5 [7.2 to 9.9] | 8.0 [6.6 to 8.9]
Statistical Analysis 1: Comparison: A: NGR-hTNF + BIC vs B: Placebo+BIC; Study with one control per experimental patient, an accrual interval of 24 months, and an additional FU after the accrual interval of 12 months.If the true HR of experimental relative to control patients was 0.726, then 195 experimental patients and 195 control patients were required to be able to reject the null hypothesis that the experimental and control survival curves were equal with probability (power)0.80 Type I error probability associated with this test of this null hypothesis was 0.05; Test type: Superiority; p = 0.58, Log Rank — The log-rank test (unstratified) was used to compare the two treatment arms. In addition, a stratified version of the log-rank test was performed with the stratification factors used for randomization; Cox regression analyses (unstratified and stratified) were performed to assess the influence of baseline covariates in an exploratory manner; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.75 to 1.18]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Defined as the time from the date of randomization until disease progression, or deathdue to any couse or the last patient was konwn to be alive. Progression is defined usind Response Evaluation Criteria In Solid Tumors Criteria (Recist v1.1), as a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition torelative increase of 20% the sum must also demonstrate an absolute increase of at least 5 mm. In addition the appearance of one or more new lesions was also considered progression
Time Frame: From the date of randomization until the date of first documented progression or date of death from any cause, wichever came first, assessed up to 48 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A: NGR-hTNF + BIC | B: Placebo+BIC
Number analyzed (Participants) | 200 | 200
months | 3.4 [2.7 to 4.1] | 3.0 [2.3 to 3.7]
Statistical Analysis 1: Comparison: A: NGR-hTNF + BIC vs B: Placebo+BIC; The log-rank test (unstratified and stratified) was used at an alpha level of 5% to test for differences in PFS between the two treatment arms. Kaplan-Meier curves and estimates were provided; Test type: Superiority; p = 0.65, Log Rank; Cox regression analyses (unstratified and stratified) was performed to assess the influence of baseline covariates in an exploratory manner; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.78 to 1.17]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate (DCR), defined as the percentage of patients who have a best-response rating of complete or partial response or stable disease, according to MPM-modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria
Time Frame: Assessed every 6-12 weeks, up to 100 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | A: NGR-hTNF + BIC | B: Placebo+BIC
Number analyzed (Participants) | 200 | 200
Participants
  Disease control rate (DCR) | 114 | 109
  Complete or partial response (CR o PR) | 3 | 6
  Stable disease (SD) | 111 | 103
  Progressive disease (PD) | 51 | 71
  Nonassessable (NA) | 35 | 20
Statistical Analysis 1: Comparison: A: NGR-hTNF + BIC vs B: Placebo+BIC; Difference in DCR between the two treatment arms were tested using a chi-squared test with 95% confidence intervals calculated in each treatment arm; Test type: Superiority; p = 0.62, Fisher Exact; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.76 to 1.68] — Logistic regression analyses were performed to assess the influence of baseline covariates in an exploratory manner

4. Secondary Outcome: Number of Partecipants With Disease Control for ≥ 6 Months
Description: Measured from the date of randomization until disease progression, or death due to any cause
Time Frame: Assessed every 6-12 weeks, up to 100 weeks
Population: Duration of disease control ≥ 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | A: NGR-hTNF + BIC | B: Placebo+BIC
Number analyzed (Participants) | 200 | 200
Participants | 84 | 76

5. Secondary Outcome: Number of Partecipants With Adverse Events
Description: All adverse events will be recorded according to CTC version 4.02 (CTC reference: http://ctep.cancer.gov/reporting/ctc.html) on the case report forms (CRFs); the investigator will decide if those events are drug related and his decision will be recorded on the forms for all adverse events.
Time Frame: Assessed every 6-12 weeks, up to 100 weeks
Population: The safety data referred to patients of both arms who received at least one treatment and is termed as safety population (n=386)
Measure: Number; unit: participants
Arm/Group | A: NGR-hTNF + BIC | B: Placebo+BIC
Number analyzed (Participants) | 193 | 193
participants
  Study-emergent AEs of any grade | 191 | 185
  Study-emergent AEs of grade 3 | 102 | 86
  Study-emergent AEs of grade 4 | 22 | 19
  Study-emergent AEs of grade 5 | 12 | 13
  Treatment-related AEs of grade 5 | 0 | 0
  Treatment discontinuation due to AEs | 31 | 24

6. Secondary Outcome: Time to LCSS Symptomatic Progression
Description: Quality of life (QoL) assessment was performed by using a questionnaire according to The Lung Cancer Symptom Scale (LCSS) . The LCSS is designed as a disease and site-specific measure of QoL particularly for use in clinical trials. It evaluates six major symptoms (loss of appetite, fatigue, cough, dyspnea, hemoptysis, and pain) associated with lung malignancies and their effect on overall symptomatic distress, functional activities, and global QoL. Within this trial the questionnaire according to LCSS was only recorded by the patient (patient's scale). QoL assessment was performed by using a questionnaire according to LCSS, which consists of nine 100-mm visual analog scales, with scores reported from 0 to 100 (0 representing the best score). The LCSS subscore is the average symptom burden index computed as the mean score for all six major symptoms. Symptomatic progression was defined as a worsening in the average symptom burden index by 25%.
Time Frame: from the date of randomization to the date of the LCSS assessment on which symptomatic progression was identified, assessed on cycle 2, cycle 4 and cycle 6 (each cycle lasted 21 days)
Population: Participants with a worsening in the average symptom burden index by 25%.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A: NGR-hTNF + BIC | B: Placebo+BIC
Number analyzed (Participants) | 175 | 185
months | 3.2 [2.1 to 4.4] | 3.0 [2.8 to 3.4]
Statistical Analysis 1: Comparison: A: NGR-hTNF + BIC vs B: Placebo+BIC; QoL assessment was performed by using a questionnaire according to LCSS, which consists of nine 100-mm visual analog scales, with scores reported from 0 to 100(the best score). The LCSS subscore is the average symptom burden index computed as the mean score for all 6 major symptoms. Symptomatic progression was defined as a worsening in the average symptom burden index by 25%; Test type: Other — Two-sided log-rank test was used to compare time to symptomatic progression between treatment arms. Median and 95% confidence limits for the time to symptomatic progression were estimated using Kaplan-Meier survival methodology. Estimates of the treatment effect were expressed as hazard ratio including 95% confidence intervals; p = 0.5806, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.68 to 1.26]

7. Secondary Outcome: Evaluation of Medical Care Utilization in the Two Treatment Arms
Description: Medical resource use data collected will be used in health economic analyses where it may be combined with other data from other sources such as cost data or other clinical parameters.
Time Frame: Assessed every 6-12 weeks, up to 100 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | A: NGR-hTNF + BIC | B: Placebo+BIC
Number analyzed (Participants) | 200 | 200
Participants
  ACE INHIBITORS, COMBINATIONS | 0 | 2
  ACE INHIBITORS, PLAIN | 5 | 2
  ADRENERGICS, INHALANTS | 7 | 10
  AMINOGLYCOSIDE ANTIBACTERIALS | 2 | 2
  ANESTHETICS, LOCAL | 0 | 4
  ANGIOTENSIN II ANTAGONISTS,COMBINATIONS | 1 | 4
  ANGIOTENSIN II ANTAGONISTS, plain | 2 | 5
  ANTACIDS | 7 | 3
  ANTERIOR PITUITARY LOBE HORMONES AND ANALOGUES | 13 | 7
  ANTIADRENERGIC AGENTS CENTRALLY ACTING | 0 | 2
  ANTIADRENERGIC AGENTS PERIPHERALLY ACTING | 0 | 2
  ANTIANDROGENS | 0 | 1
  ANTIARRHYTHMICS, CLASS I AND III | 4 | 3
  ANTIBIOTICS FOR TOPICAL USE | 0 | 4
  ANTIDEPRESSANTS | 17 | 2
  ANTIDIARRHEAL MICROORGANISMS | 2 | 1
  ANTIEMETICS AND ANTINAUSEANTS | 107 | 110
  ANTIEPILEPTICS | 3 | 2
  ANTIFIBRINOLYTICS | 1 | 0
  ANTIFUNGALS FOR TOPICAL USE | 2 | 0
  ANTIGLAUCOMA PREPARATIONS AND MIOTICS | 0 | 1
  ANTIGOUT PREPARATIONS | 10 | 12
  ANTIHISTAMINES FOR SYSTEMIC USE | 66 | 31
  ANTIINFECTIVES | 0 | 1
  ANTIINFLAMMATORY AGENTS AND ANTIINFECTIVES IN COM | 0 | 2
  ANTIINFLAMMATORY ANANTIRHEUMATIC PRODUCTSD | 58 | 65
  ANTIMETABOLITES | 1 | 1
  ANTIMYCOTICS FOR SYSTEMIC USE | 15 | 14
  ANTIPROPULSIVES | 4 | 8
  ANTIPRURITICS | 3 | 2
  ANTIPSYCHOTICS | 7 | 3
  ANTITHROMBOTIC AGENTS | 41 | 42
  ANTIVERTIGO PREPARATIONS | 2 | 1
  ANXIOLYTICS | 24 | 16
  ASCORBIC ACID (VITAMIN C) | 0 | 1
  BACTERIAL VACCINES | 1 | 0
  BELLADONNA AND DERIVATIVES | 3 | 4
  BETA BLOCKING AGENTS AND OTHER ANTIHYPERTENSIVES | 11 | 15
  BETA-LACTAM ANTIBACTERIALS, PENICILLINS | 38 | 29
  BILE THERAPY | 1 | 1
  BLOOD AND RELATED PRODUCTS | 21 | 26
  BLOOD GLUCOSE LOWERING DRUGS EXCL. INSULINS | 2 | 6
  CALCIUM | 19 | 12
  CAPILLARY STABILIZING | 1 | 0
  CARDIAC GLYCOSIDES | 1 | 3
  CARDIAC STIMULANTS EXCL CARDIAC GLYCOSIDES | 1 | 0
  CORTICOSTEROIDS FOR SYSTEMIC USE, PLAIN | 138 | 108
  CORTICOSTEROIDS, PLAIN | 2 | 1
  COUGH SUPPRESSANTS AND EXPECTORANTS, COMBINATIONS | 2 | 5
  COUGH SUPPRESSANTS, EXCL. COMBINATIONS WITH EXPEC | 7 | 17
  DECONGESTANTS AND ANTIALLERGICS | 0 | 1
  DIRECT ACTING ANTIVIRALS | 2 | 2
  DIURETICS AND POTASSIUM-SPARING AGENTS | 6 | 3
  DRUGS AFFECTING BONE | 2 | 3
  DRUGS FOR CONSTIPATION | 39 | 63
  DRUGS FOR FUNCTIONAL GASTROINTESTINAL DISORDERS | 3 | 5
  DRUGS FOR PEPTIC ULCER AND GASTRO-OESOPHAGEAL REF | 74 | 71
  DRUGS FOR TREATMENT OF TUBERCULOSIS | 2 | 0
  DRUGS USED IN BENIGN PROSTATIC HYPERTROPHY | 4 | 1
  ECTOPARASITICIDES, INC SCABICIDESL. | 0 | 1
  EMOLLIENTS AND PROTECTIVES | 1 | 0
  EXPECTORANTS EXCL COMBINATIONS WITH COUGH SUPPR. | 14 | 9
  HIGH-CEILING DIURETICS | 19 | 20
  HORMONES AND RELATED AGENTS | 0 | 1
  HYPNOTICS AND SEDATIVES | 14 | 14
  HYPOTHALAMIC HORMONES | 0 | 1
  I.V. SOLUTION ADDITIVES | 17 | 21
  I.V. SOLUTIONS | 6 | 10
  IMMUNOSTIMULANTS | 20 | 19
  INSULINS AND ANALOGUES | 5 | 0
  INTESTINAL ANTIINFECTIVES | 3 | 2
  IRON PREPARATIONS | 14 | 9
  LIPID MODIFYING AGENTS, PLAIN | 4 | 4
  LOW-CEILING DIURETICS, EXCL THIAZIDES | 1 | 0
  MACROLIDES, LINCOSAMIDES AND STREPTOGRAMINS | 8 | 14
  MULTIVITAMINS, COMBINATIONS | 1 | 4
  MULTIVITAMINS, PLAIN | 4 | 5
  MUSCLE RELAXANTS, CENTRALLY ACTING AGENTS | 0 | 1
  MYDRIATICS AND CYCLOPLEGICS | 2 | 3
  OPIOIDS | 135 | 160
  OTHER ANALGESICS AND ANTIPYRETICSD | 105 | 93
  OTHER ANTIANEMIC PREPARATIONS | 20 | 20
  OTHER ANTIBACTERIALS | 4 | 5
  OTHER ANTIDIARRHEALS | 1 | 0
  OTHER ANTINEOPLASTIC AGENTS | 0 | 2
  OTHER BETA-LACTAM ANTIBACTERIALS | 8 | 9
  OTHER CARDIAC PREPARATIONS | 3 | 0
  OTHER DRUGS FOR ACID RELATED DISORDERS | 0 | 1
  OTHER DRUGS FOR OBSTRUCTIVE | 7 | 8
  OTHER MINERAL SUPPLEMENTS | 4 | 5
  OTHER NUTRIENTS | 4 | 7
  OTHER OPHTHALMOLOGICALS | 0 | 1
  OTHER PLAIN VITAMIN PREPARATIONS | 2 | 0
  OTHER RESPIRATORY SYSTEM PRODUCTS | 2 | 0
  OTHER SYSTEMIC DRUGS FOR OBSTRUCTIVE AIRWAY DISEA | 3 | 1
  OTHER VITAMIN PRODUCTS, COMBINATIONS | 1 | 2
  PERIPHERAL VASODILATORS | 0 | 1
  POTASSIUM | 4 | 5
  POTASSIUM-SPARING AGENTS | 1 | 5
  PROPULSIVES | 68 | 87
  PSYCHOLEPTICS AND PSYCHOANALEPTICS | 0 | 1
  PSYCHOSTIMULANTS, | 0 | 1
  QUINOLONE ANTIBACTERIALS | 31 | 36
  SELECTIVE CALCIUM CHANNEL BLOCKERS WITH MAINLY VA | 1 | 6
  STOMATOLOGICAL PREPARATIONS | 20 | 19
  SULFONAMIDES AND TRIMETHOPRIM | 2 | 0
  TETRACYCLINES | 0 | 4
  THYROID PREPARATIONS | 2 | 0
  TOPICAL PRODUCTS FOR JOINT AND MUSCULAR PAIN | 1 | 2
  UROLOGICALS | 3 | 1
  VASODILATORS USED IN CARDIAC DISEASES | 0 | 2
  VIRAL VACCINES | 1 | 0
  VITAMIN A AND D | 0 | 5
  VITAMIN B1, PLAIN AND IN COMBINATION WITH VITAMIN | 0 | 3
  VITAMIN B12 AND FOLIC ACID | 7 | 11
  VITAMIN K AND OTHER HEMOSTATICS | 1 | 3
  SELECTIVE CALCIUM CHANNEL BLOCKERS WITH DIRECT CA | 3 | 4

ADVERSE EVENTS:
Time Frame: Through study completation, an average of 2 years
Arm/Group | A: NGR-hTNF + BIC | B: Placebo+BIC
All-Cause Mortality (participants affected / at risk) | 12/193 | 13/193
Serious Adverse Events (participants affected / at risk) | 56/193 | 54/193
Other Adverse Events (participants affected / at risk) | 190/193 | 185/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: NGR-hTNF + BIC (N=193) | B: Placebo+BIC (N=193)
Paraneoplastic fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain mets (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain mets (Immune system disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Mucositis (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 (2) | 2 (2)
Death (General disorders) | 3 (3) | 2 (2)
Hyperpyrexia (General disorders) | 1 | 0
Ischaemic ulcer to left heel (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 3 (3) | 3 (3)
Deterioration of clinical status (General disorders) | 1 (1) | 1 (1)
Admitted for pain control (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Uncertain study medication dose delivered (Injury, poisoning and procedural complications) | 4 (4) | 9 (9)
Drug infusion reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Occipital trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infection (chest) with normal ANC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenic fever (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Superior sagittal sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Right hemispheric cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abnormal renal function (Renal and urinary disorders) | 1 (1) | 0 (0)
Pain right chest wall + right shoulder (Musculoskeletal and connective tissue disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 1 (1)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Infection - source unknown (Infections and infestations) | 1 (1) | 0 (0)
Viral gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac arresr (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 | 0
Condition aggraveted (General disorders) | 4 (4) | 5 (5)
Lower Respiratory Tract Infection (Infections and infestations) | 2 (2) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1)
. Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Pleural Mesothelioma (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Jacksonian seizure (Nervous system disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: NGR-hTNF + BIC (N=193) | B: Placebo+BIC (N=193)
Hypertension (Vascular disorders) | 12 (16) | 12 (15)
Hypotension (Vascular disorders) | 10 (12) | 7 (9)
Neutropenia (Blood and lymphatic system disorders) | 57 (162) | 60 (119)
Anaemia (Blood and lymphatic system disorders) | 34 (58) | 42 (79)
Thrombocytopenia (Blood and lymphatic system disorders) | 26 (56) | 23 (47)
Leukopenia (Blood and lymphatic system disorders) | 24 (85) | 20 (24)
Dysponoea (Respiratory, thoracic and mediastinal disorders) | 63 (94) | 56 (80)
Cough (Respiratory, thoracic and mediastinal disorders) | 39 (59) | 47 (71)
Dizziness (Nervous system disorders) | 11 (12) | 12 (14)
Dysgeusia (Nervous system disorders) | 10 (10) | 6 (7)
Headache (Nervous system disorders) | 15 (16) | 13 (15)
Pheripheral neuropathy (Nervous system disorders) | 12 (20) | 12 (15)
Chills (General disorders) | 104 (462) | 23 (29)
Fatigue (General disorders) | 93 (166) | 94 (180)
Pain (General disorders) | 91 (179) | 89 (184)
Pyrexia (General disorders) | 48 (103) | 39 (67)
Oedema (General disorders) | 26 (31) | 25 (29)
Mucosal inflammation (General disorders) | 20 (29) | 17 (23)
Insomnia (Psychiatric disorders) | 11 (12) | 12 (12)
Nausea (Gastrointestinal disorders) | 61 (122) | 62 (130)
Constipation (Gastrointestinal disorders) | 42 (65) | 45 (65)
Vomiting (Gastrointestinal disorders) | 33 (61) | 38 (81)
Diarrhoea (Gastrointestinal disorders) | 20 (39) | 36 (58)
Dyspepsia (Gastrointestinal disorders) | 10 (12) | 11 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (12) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (15) | 8 (8)
Decreased appetite (Metabolism and nutrition disorders) | 46 (68) | 51 (76)
Hypocalcaemia (Metabolism and nutrition disorders) | 12 (21) | 5 (6)
Respiratory tract infection (Infections and infestations) | 13 (15) | 10 (13)
Transaminases Increased (Investigations) | 14 (37) | 7 (20)
Abdominal disconfort (Gastrointestinal disorders) | 1 (1) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes